CLINICAL TRIAL: NCT05548101
Title: Prospective, Randomized Trial Comparing ICSI to Insemination for Non-Male Factor Patients Undergoing PGT-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Fertility Center (Other)
Collaborators: Ovation Fertility (Other)
Responsible Party: Principal Investigator, Kaylen Silverberg MD, MD, Texas Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICSI
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Infertility
Keywords: Infertility; ICSI; Intracytoplasmic Sperm Injection; non-male factor infertility; IVF; In Vitro Fertilization; PGT-A
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled clinical trial
Who Masked: Participant
Masking Description: Patient will be blinded to use of ICSI versus conventional insemination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Insemination (No Intervention): Oocytes will be fertilized via conventional insemination: Oocytes will be washed with multipurpose handling medium (MHM) plus 0.5% human serum albumin (HSA). Excess cumulus cells and blood will be trimmed. Oocytes will be transferred to a dish containing Irvine Scientific Continuous Cell Culture Complete Medium with two oocytes per dish. The dish will then be transferred to the incubator. Insemination will occur 4-6 hours post-retrieval. Sperm will be collected as a fresh specimen and washed with Irvine Scientific Continuous Single Culture-NX. Sperm concentration and motility will be assessed before and after washing according to WHO 6th edition criteria. Sperm will be prepared to achieve a concentration of 200,000 sperm per 100 microliter drop. 6 drops of prepared sperm will be added to each dish.
- Intracytoplasmic Sperm Injection (ICSI) (Active Comparator): Oocytes will be fertilized via ICSI: Oocytes will be washed with multipurpose handling medium (MHM) plus 0.5% human serum albumin (HSA). Excess cumulus cells and blood will be trimmed. Oocytes will be transferred to a dish containing Irvine Scientific Continuous Cell Culture Complete Medium with two oocytes per dish. The dish will then be transferred to the incubator. Oocytes will be immediately exposed to hyaluronidase to strip the cumulus and coronal cells. Embryologists will assess the maturation status under inverted microscopy. ICSI will be performed on all mature metaphase II oocytes 4 hours after retrieval. Injected oocytes will then be placed in a fresh culture dish and returned to the incubator.
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — Using the injecting pipet, one sperm will be isolated. Using the tip of the injecting pipet, the sperm tail will be broken by trapping it between the pipet and bottom of the dish. The sperm will be picked up in the pipet. The oocyte will be positioned so the polar body is at the 12 o'clock or 6 o'clock position. The sperm injecting pipet will be positioned at the 3 o'clock position of the oocyte. The injecting pipet will be advanced into the oocyte cytoplasm and the cytoplasm will be gently aspirated until the oocyte membrane breaks. The sperm will then be injected into the cytoplasm of the oocyte. The pipet will then be withdrawn from the oocyte.
  Other Names: Intracytoplasmic Sperm Injection
  Arms: Intracytoplasmic Sperm Injection (ICSI)

SUMMARY:
Intracytoplasmic sperm injection (ICSI) is a procedure performed during in vitro fertilization (IVF) in which a single sperm is injected directly into an oocyte. This procedure was developed for male factor infertility due to its requirement for a very small number of viable sperm. However, its use has expanded and is now recommended for IVF cycles in which preimplantation genetic testing for aneuploidies (PGT-A) is performed on blastocysts. We hypothesize that the ICSI procedure may interfere with the normal meiosis II process that occurs during fertilization, and lead to a higher rate of aneuploid blastocysts. In our study we will randomly assign non-male factor infertility patients to either conventional insemination or ICSI and compare the rate of karyotypically normal embryos in each group.

DETAILED DESCRIPTION:
Intracytoplasmic sperm injection (ICSI) is a procedure performed during in vitro fertilization (IVF) in which a single sperm is injected directly into an oocyte. This procedure was developed for male factor infertility due to its requirement for a very small number of viable sperm. Fertilization rates have been noted to be approximately 60-70%, comparable to traditional insemination. Its use has expanded and is now recommended for IVF cycles in which preimplantation genetic testing for aneuploidies (PGT-A) is performed on blastocysts. With PGT-A, euploid embryos can be selected to transfer, ultimately increasing implantation rates, raising ongoing pregnancy rates, and reducing the incidence of miscarriage. The recommendation to utilize ICSI for all PGT-A cycles was initially based on ensuring monospermic fertilization and minimizing contamination from additional sperm attached to the oocyte's zona pellucida during the use of polymerase chain reaction (PCR) for genetic testing. However, this is of less concern with newer next generation sequencing molecular techniques that are now used and enable much higher resolution analysis.

It has been suggested that ICSI may slightly increase the risk of imprinting disorders and birth defects, and significantly increases the cost of IVF. Meiosis II occurs during oocyte fertilization, and as such, any disruption of the meiosis apparatus could potentially lead to errors in chromosomal division. We hypothesize that the ICSI procedure may interfere with the normal meiosis process and lead to a higher rate of aneuploid blastocysts.

Our study will randomly assign patients with non-male factor infertility undergoing IVF with PGT-A at Texas Fertility Center to either conventional insemination or ICSI. Women aged 18-39 years old with at least 10 oocytes following retrieval will be included. Initial semen analysis must have greater than or equal to 16 million sperm/mL, 42% motile sperm, 16.4 million total motile sperm, 30% progressive motility, and 4% normal morphology (as defined by WHO 6th edition). Patients will be excluded for any of the following: any fertilization failure or more than one implantation failure from previous IVF cycles; male factor infertility as defined by sperm concentration less than 16 million sperm/mL, motility less than 42%, total motile count less than 16.4 million, progressive motility less than 30%, and normal morphology less than 4%; female partner over age 39 years old; 9 or fewer oocytes following retrieval; couples requiring single gene analysis by preimplantation genetic testing for monogenic disorders (PGT-M); ICSI for any reason other than PGT-A.

The female partner will undergo controlled ovarian stimulation with a protocol chosen by each patient's physician based on patient age, history, and ovarian reserve. Recombinant follicle stimulating hormone (FSH) (Gonal F or Follistim) and human menopausal gonadotropin (Menopur) will be used for stimulation. Gonadotropin-releasing hormone (GnRH) agonist (Lupron) or antagonist (Cetrotide or Ganirelix) with or without oral contraceptive pills (OCPs) or with estradiol priming will be used for suppression of ovulation. The patient will be monitored every 1-3 days utilizing ultrasound to measure follicular growth as well as blood estradiol levels, with medication and dosing adjusted accordingly. Oocyte maturation will be triggered with gonadotropin-releasing hormone (GnRH) agonist (Lupron) and/or human chorionic gonadotropin (Novarel or Pregnyl). Oocyte retrieval will occur 36 hours after trigger according to standard protocols at our center.

Oocytes will be washed with multipurpose handling medium (MHM) plus 0.5% human serum albumin (HSA). Excess cumulus cells and blood will be trimmed. Oocytes will be transferred to a dish containing Irvine Scientific Continuous Cell Culture Complete Medium with two oocytes per dish. The dish will then be transferred to the incubator.

Oocytes designated for ICSI will be immediately exposed to hyaluronidase to strip the cumulus and coronal cells. Embryologists will assess the maturation status under inverted microscopy. ICSI will be performed on all mature metaphase II oocytes 4 hours after retrieval. Injected oocytes will then be placed in a fresh culture dish and returned to the incubator.

For oocytes designated for conventional insemination, insemination will occur 4-6 hours post-retrieval. Sperm will be collected as a fresh specimen and washed with Irvine Scientific Continuous Single Culture-NX. Sperm concentration and motility will be assessed before and after washing according to WHO 6th edition criteria. Sperm will be prepared to achieve a concentration of 200,000 sperm per 100 microliter drop. 6 drops of prepared sperm will be added to each dish.

The following morning after ICSI or conventional insemination (Day 1), oocytes will be examined for fertilization. Zygotes with two pronuclei (2PN) will be kept in group culture to be assessed again on Days 5, 6, and 7. Embryos that reach the blastocyst stage will be morphologically graded by our embryologists. The Inner Cell Mass (ICM) and trophectoderm will each be given a grade of Good (G), Fair (F), or Poor (P). Blastocysts with grades G or F will undergo trophectoderm biopsy and subsequent vitrification. Trophectoderm biopsy will be performed using a standard protocol: Hatching trophoblast cells opposite the inner cell mass will be gently aspirated into the biopsy pipet. The SaturnActive laser will be used to separate 3-5 cells. Biopsied cells will be prepared and loaded in PCR tubes according to the PGT-A center protocols and stored at -20 degrees Celsius until transportation to the testing center.

Next Generation Sequencing will be used to analyze samples at a PGT testing center (Ovation Genetics, Cooper Genomics, Natera, RGI, or Genomic Prediction). Copy number variations will be used to diagnose ploidy status. Euploidy will be defined as a normal number of chromosomes. Aneuploidy will be defined as an abnormal number of chromosomes. Mosaicism will be defined as 30-70% mosaicism, whereas less than 30% mosaicism will be considered euploidy, and greater than 70% mosaicism will be considered aneuploidy. PGT-A outcomes will be analyzed for percentage of euploid, aneuploid, mosaic, and no result embryos.

ELIGIBILITY:
Inclusion Criteria:

* Female partner aged 18-39 years old with at least 10 oocytes following retrieval
* Male partner with initial semen analysis with greater than or equal to 16 million sperm/mL, greater than or equal to 42% motile sperm, greater than or equal to 16.4 million total motile sperm, greater than or equal to 30% progressive motility, and greater than or equal to 4% normal morphology (as defined by WHO 6th edition)

Exclusion Criteria:

* Fertilization failure or more than one implantation failure from previous IVF cycles
* Male factor infertility as defined by sperm concentration less than 16 million sperm/mL, motility less than 42%, total motile count less than 16.4 million, progressive motility less than 30%, or normal morphology less than 4%
* Female partner over age 39 years old
* Female partner with 9 or fewer oocytes following retrieval
* Singe gene analysis by preimplantation genetic testing for monogenic disorders (PGT-M) being performed
* ICSI being performed for any reason other than PGT-A

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — There must be a female partner to undergo oocyte retrieval and a male partner to provide sperm for insemination.
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of karyotypically normal blastocysts | 2 weeks after oocyte retrieval
  Aneuploidy will be defined as an abnormal number of chromosomes. Mosaicism will be defined as 30-70% mosaicism, whereas less than 30% mosaicism will be considered euploidy, and greater than 70% mosaicism will be considered aneuploidy. PGT-A outcomes will be analyzed for percentage of euploid, aneuploid, mosaic, and no result embryos. Rate of karyotypically normal blastocysts will be defined as the number of euploid blastocysts divided by the number of normally fertilized (2PN) embryos in that group. We will also assess the number of euploid embryos as a percentage of the total number of inseminated or injected oocytes.

SECONDARY OUTCOMES:
Rate of blastocyst development | 1 week after oocyte retrieval
  Embryos that reach the blastocyst stage will be morphologically graded by our embryologists. The Inner Cell Mass (ICM) and trophectoderm will each be given a grade of Good (G), Fair (F), or Poor (P). Blastocysts with both grades G or F will undergo trophectoderm biopsy and subsequently vitrified. We will assess the rate of development by dividing the number of freeze quality blastocysts by the total number of inseminated or injected oocytes. We will also assess the number of freeze quality embryos as a percentage of 2PN embryos per group.
Fertilization rate | 1 day after oocyte retrieval
  The following morning after ICSI or conventional insemination (Day 1), oocytes will be examined for fertilization. Zygotes with two pronuclei (2PN) will be kept in group culture to be assessed again on Days 5, 6, and 7. We will assess the percentage of total retrieved oocytes that were fertilized with each type of insemination.

CONTACTS AND LOCATIONS:
Overall Officials: Kaylen Silverberg, MD, Principal Investigator — Texas Fertility Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. Electronic address: asrm@asrm.org. Intracytoplasmic sperm injection (ICSI) for non-male factor indications: a committee opinion. Fertil Steril. 2020 Aug;114(2):239-245. doi: 10.1016/j.fertnstert.2020.05.032. Epub 2020 Jul 9. PMID 32654822
- [Background] Palmerola KL, Vitez SF, Amrane S, Fischer CP, Forman EJ. Minimizing mosaicism: assessing the impact of fertilization method on rate of mosaicism after next-generation sequencing (NGS) preimplantation genetic testing for aneuploidy (PGT-A). J Assist Reprod Genet. 2019 Jan;36(1):153-157. doi: 10.1007/s10815-018-1347-6. Epub 2018 Oct 25. PMID 30362056
- [Background] Niu X, Long J, Gong F, Wang W. Does ICSI for in vitro fertilization cause more aneuploid embryos? Mol Cytogenet. 2020 Jul 1;13:27. doi: 10.1186/s13039-020-00497-z. eCollection 2020. PMID 32636925
- [Background] Swearman HK, Liperis G, Crittlendon J, Sjoblom C. Fertilization by ICSI results in significantly higher aneuploidy rates compared to IVF, in embryos analysed by next generation sequencing (NGS) or comparative genome hybridization (CGH) array. ASRM Poster Session Volume 110, Issue 4, Supplement, E346-347. 2018 Sep.
- [Background] Deng J, Kuyoro O, Zhao Q, Behr B, Lathi RB. Comparison of aneuploidy rates between conventional in vitro fertilization and intracytoplasmic sperm injection in in vitro fertilization-intracytoplasmic sperm injection split insemination cycles. F S Rep. 2020 Jul 27;1(3):277-281. doi: 10.1016/j.xfre.2020.07.006. eCollection 2020 Dec. PMID 34223256
- [Background] Kandil H, Agarwal A, Saleh R, Boitrelle F, Arafa M, Vogiatzi P, Henkel R, Zini A, Shah R. Editorial Commentary on Draft of World Health Organization Sixth Edition Laboratory Manual for the Examination and Processing of Human Semen. World J Mens Health. 2021 Oct;39(4):577-580. doi: 10.5534/wjmh.210074. Epub 2021 Jun 11. No abstract available. PMID 34169684